CLINICAL TRIAL: NCT05702216
Title: Étude de Non-infériorité d'un Programme de télé-réadaptation Cardiovasculaire Sous Une Forme Hybride Par Rapport à Une rééducation réadaptation Cardiovasculaire Classique
Brief Title: Non-inferiority Study of a Cardiac Tele-rehabilitation in Hybrid Form Compared to a Cardiac Rehabilitation
Acronym: TELEREHAB
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Clinique de la Mitterie (Other)
Responsible Party: Principal Investigator, Michaël RACODON, clinical research coordinator, Clinique de la Mitterie
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: N° 2021-A03116-35
Record Dates: First submitted 2023-01-18; First posted 2023-01-27 (Actual); Last update posted 2023-12-27 (Actual); Status verified 2023-12

CONDITIONS: Cardiac Tele-rehabilitation
Keywords: Cardiac tele-rehabilitation, cardiac rehabilitation
MeSH Terms: interventions — Rehabilitation

STUDY DESIGN:
Intervention Model Description: Randomization in two groups: a Hybrid Tele-pulmonary Rehabilitation group and a classic Rehabilitation group.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cardiac rehabilitation (Other)
  Interventions: Other: Rehabilitation
- Cardiac Tele-rehabilitation (Other): Tele cardiac rehabilitation in hybrid form
  Interventions: Other: Rehabilitation

INTERVENTIONS:
Other: Rehabilitation — Hybrid approach in cardiac telerehabilitation. Patients underwent 20 cardiac rehabilitation sessions: alternatively, patients underwent 10 classical cardiac rehabilitation sessions in the clinic and 10 cardiac telerehabilitation sessions at home.

SUMMARY:
Cardiac tele-rehabilitation in a hybrid form can be a choise for the management of cardiovascular diseases. The aim is to increase the participation rate of patients in cardiac rehabilitation.

This new form of care can be as effective as traditional care.

DETAILED DESCRIPTION:
The Covid-19 pandemic has had indirect effects on the health system, particularly in the management of cardiovascular diseases. Rehabilitation centres had to adapt their operation to the recommendations of health authorities. The choice appeared to be unavoidable: tele-rehabilitation care in a hybrid form. Moreover, Many patients do not participate at this kind of care. Many identified factors can explain this low rate of participation : a lack of proximity facilities does not promote patient participation.

The objective of this study is to demonstrate a comparable effectiveness between a cardiac telerehabilitation programme in hybrid form and a cardiac classic rehabilitation programme.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 ans
* Patients with heart disease
* Inclusion in the rehabilitation program

Exclusion Criteria:

* Cardiac decompensation
* No stabilised acute coronary syndrome
* Decompensated heart failure
* Severe ventricular rhythm disorders
* Severe functional limitation

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2021-10-29 (Actual); Primary Completion 2022-09-05 (Actual); Study Completion 2023-03-31 (Actual)

PRIMARY OUTCOMES:
6-minute walk test | 6 weeks before baseline
  Distance covered in the 6-minute walk test

SECONDARY OUTCOMES:
Stress test | 6 weeks before baseline
  12-lead electrocardiogram
Wall Squat Test | 6 weeks before baseline
  Muscular endurance

CONTACTS AND LOCATIONS:
Overall Officials: Michaël RACODON, Ph.D, Study Director — CLINIQUE LA MITTERIE
Locations (1):
- Clinique la Mitterie, Lille, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Racodon M, Peze T, Masson P. Analysis of physical exercise in cardiac patients following cardiovascular rehabilitation. Acta Cardiol. 2020 Nov;75(7):598-603. doi: 10.1080/00015385.2019.1639269. Epub 2019 Jul 17. PMID 31314680